CLINICAL TRIAL: NCT00332592
Title: Intragastric and Intraperitoneal Microdialysis in Infants With NEC
Brief Title: Intragastric and Peritoneal Microdialysis in Infants With Necrotizing Enterocolitis (NEC)
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Niels Qvist, Surgical department A, Odense University Hospital
Other Study IDs: VF-20060037
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-05

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing Enterocolitis; Intragastric microdialysis; Peritoneal microdialysis; Infants
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
NEC is a serious inflammatory bowel disease, which almost only strikes infants with low birth weight and low gestational age. The morbidity and mortality rates are high, and early diagnosis and treatment is mandatory. The primary aim of the present study is to investigate the clinical use of intragastric microdialysis and whether it is able to select patients, who may benefit from either medical or surgical therapy. The aim of intraperitoneal microdialysis is to evaluate whether changes in intraperitoneal microdialysis reflect the clinical outcome after laparotomy.

DETAILED DESCRIPTION:
Neonates who are hospitalized because of suspicion of NEC are subjected to intragastric microdialysis during the observation period. The catheter is placed in the stomach via the naso-oesophageal route. If surgery is necessary a microdialysis catheter is placed in the peritoneal cavity prior to wound closure. Samples are collected every 4-hour. Samples will be analyzed continuously but the results will not be included in the clinical evaluation of the patient.

A total of 20 patients will be included in this pilot study. The results of the intragastric and peritoneal microdialysis will be compared with the clinical course, s-lactate, radiological and pathological findings in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who are hospitalized because of suspicion of NEC.
* Neonates who has surgery because of NEC.

Exclusion Criteria:

* Non-acceptance from the child's parents or custody holder

Ages: 3 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature children with NEC
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Surgical department A, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Pedersen ME, Dahl M, Qvist N. Intraperitoneal microdialysis in the postoperative surveillance after surgery for necrotizing enterocolitis: a preliminary report. J Pediatr Surg. 2011 Feb;46(2):352-6. doi: 10.1016/j.jpedsurg.2010.11.015. PMID 21292087